CLINICAL TRIAL: NCT02897570
Title: Effect of Glucose Versus Mixed Breakfast on Metabolic and Neurofunctional Responses in Healthy Individuals
Brief Title: Metabolic and Neurofunctional Responses to Breakfasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Collaborators: Soremartec Italia S.r.l. (Unknown)
Responsible Party: Principal Investigator, Anna Ferrulli, MD, Ospedale San Donato
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Colazioni/4
Record Dates: First submitted 2016-08-26; First posted 2016-09-13 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Feeding Behaviors; Lack of Satiety; Attention Deficit and Disruptive Behavior Disorders
Keywords: ghrelin; breakfast meal; P-300
MeSH Terms: conditions — Feeding Behavior; Attention Deficit and Disruptive Behavior Disorders | interventions — Glucose; Milk; Edible Grain; Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glucose (Active Comparator): EEG_pre + Oral glucose tolerance test (50-g OGTT) + EEG_post
  Interventions: Dietary Supplement: Glucose; Device: EEG_pre; Device: EEG_post
- Milk + Cereals (Experimental): EEG_pre + B1: milk (125ml) and cereals (30g) + EEG_post
  Interventions: Dietary Supplement: Milk & Cereals; Dietary Supplement: Milk, apple & snack; Device: EEG_pre; Device: EEG_post
- Milk + Apple + Snack (Experimental): EEG_pre + B2: milk (220ml), apple (200g) and cream chocolate filled sponge cake (30g) + EEG_post
  Interventions: Dietary Supplement: Milk & Cereals; Dietary Supplement: Milk, apple & bread w/ cream; Device: EEG_pre; Device: EEG_post
- Milk + Apple + Bread w/ cream (Experimental): EEG_pre + B3: milk (125ml), apple (150g), and bread (50g) with hazelnut chocolate cream (15g) + EEG_post
  Interventions: Dietary Supplement: Milk & Cereals; Dietary Supplement: Milk, apple & bread w/ cream; Device: EEG_pre; Device: EEG_post

INTERVENTIONS:
Dietary Supplement: Glucose — 50g of glucose dissolved in 250 to 300ml of water was drunk. Prior and upon completion of each glucose tolerance test, an EEG was performed.
  Arms: Glucose
Dietary Supplement: Milk & Cereals — A breakfast (B1) including a glass of milk (125ml) and 30 g-corn flakes was consumed. Prior and upon completion of each tolerance test, an EEG was performed
  Arms: Milk + Apple + Bread w/ cream; Milk + Apple + Snack; Milk + Cereals
Dietary Supplement: Milk, apple & snack — A breakfast (B2) including a glass of milk (220ml), an apple (200g), a cream chocolate filled sponge cake (30g) was consumed. Prior and upon completion of each meal tolerance test, an EEG was performed.
  Arms: Milk + Cereals
Dietary Supplement: Milk, apple & bread w/ cream — A breakfast (B3) including a glass of milk (125ml), an apple (150g), bread (50g, hazelnut chocolate cream (15g) was consumed. Prior and upon completion of each meal tolerance test, an EEG was performed.
  Arms: Milk + Apple + Bread w/ cream; Milk + Apple + Snack
Device: EEG_pre — Electroencephalography (EEG) was performed prior each tolerance test to assess frontal P300-evoked potentials
Device: EEG_post — Electroencephalography (EEG) was performed upon completion of each tolerance test to assess frontal P300-evoked potentials

SUMMARY:
This study aims at assessing the effects of glucose and different types of breakfast on metabolic and neurofunctional responses in healthy individuals.

Twelve healthy subjects, on a stable diet, in a randomized-crossover fashion, received either a 50 g glucose load (control) or one of these breakfast:

B1: milk (125ml) and cereals (30g); B2: milk (220ml), apple (200g) and cream chocolate filled sponge cake (30g); B3: milk (125ml), bread (50g), apple (150g) and hazelnut cream chocolate (15g). Prior and upon completion of each tolerance test, an EEG was performed to measure frontal P300-evoked potentials.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 24.9 kg/m2
* normal glucose tolerance
* stable diet

Exclusion Criteria:

* type 1 and type 2 diabetes
* impaired glucose tolerance
* dyslipidemia
* metabolic syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of glucose vs different kind of breakfasts on cognitive performances via brain evoked-potentials measure | The incremental (post-pre) frontal P300 potential was assessed as a "change" ( before and 180 min after consumption)
  On the same morning of the glucose tolerance test, before and 180 min after consumption, an EEG was performed to record P300 wave-evoked potentials.

SECONDARY OUTCOMES:
Effect of glucose vs different kind of breakfasts on AUC_glycemia in healthy subjects | Blood samples are drawn at -15, 0, 15, 30, 45, 60, 75, 90, 120 minutes with respect to the ingestion.
  The incremental area under plasma glucose concentration curve (AUC_glycemia) was used as summary measures of the metabolic responses resulting from the intake of either glucose or one of the 3 breakfasts. The incremental AUC was calculated as the difference between the total AUC and the product of the basal, pre-test concentration time during the experiment (i.e., 120 min).
Effect of glucose vs different kind of breakfasts on AUC_ghrelinemia in healthy subjects. | Blood samples are drawn at -15, 0, 15, 30, 45, 60, 75, 90, 120 minutes with respect to the ingestion.
  The incremental area under plasma ghrelin concentration curve (AUC_ghrelinemia) was used as summary measures of the metabolic responses resulting from the intake of either glucose or one of the 3 breakfasts. The incremental AUC was calculated as the difference between the total AUC and the product of the basal, pre-test concentration time during the experiment (i.e., 120 min).
Effect of glucose vs different kind of breakfasts on AUC_insulinemia in healthy subjects. | Blood samples are drawn at -15, 0, 15, 30, 45, 60, 75, 90, 120 minutes with respect to the ingestion.
  The incremental area under plasma insulim concentration curve (AUC_insulinemia) was used as summary measures of the metabolic responses resulting from the intake of either glucose or one of the 3 breakfasts. The incremental AUC was calculated as the difference between the total AUC and the product of the basal, pre-test concentration time during the experiment (i.e., 120 min).

CONTACTS AND LOCATIONS:
Locations (1):
- San Donato Hospital, San Donato Milanese, MI, Italy

REFERENCES:
- [Background] Barclay AW, Brand-Miller JC, Wolever TM. Glycemic index, glycemic load, and glycemic response are not the same. Diabetes Care. 2005 Jul;28(7):1839-40. doi: 10.2337/diacare.28.7.1839. No abstract available. PMID 15983358
- [Background] Franz MJ. The glycemic index: not the most effective nutrition therapy intervention. Diabetes Care. 2003 Aug;26(8):2466-8. doi: 10.2337/diacare.26.8.2466. No abstract available. PMID 12882880
- [Background] Esposito K, Giugliano D. Low-glycemic load diet and resting energy expenditure. JAMA. 2005 Mar 9;293(10):1189; auhor reply 1189-90. doi: 10.1001/jama.293.10.1189-a. No abstract available. PMID 15755939
- [Background] Benedini S, Codella R, Caumo A, Marangoni F, Luzi L. Different circulating ghrelin responses to isoglucidic snack food in healthy individuals. Horm Metab Res. 2011 Feb;43(2):135-40. doi: 10.1055/s-0030-1269900. Epub 2011 Jan 10. PMID 21225542
- [Background] Cummings DE, Purnell JQ, Frayo RS, Schmidova K, Wisse BE, Weigle DS. A preprandial rise in plasma ghrelin levels suggests a role in meal initiation in humans. Diabetes. 2001 Aug;50(8):1714-9. doi: 10.2337/diabetes.50.8.1714. PMID 11473029